CLINICAL TRIAL: NCT01195233
Title: Comparison Study of BioXtra Spray and Mouth Rinse in Patient With Radiation-induced Xerostomia
Brief Title: Comparative Analysis of BioXtra on Xerostomia
Acronym: BioXtra
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Collaborators: Imam Khomeini Hospital (Other)
Responsible Party: Dr Mahin Bakhshi, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: QUMS 1350
Record Dates: First submitted 2010-08-27; First posted 2010-09-06 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2010-07

CONDITIONS: Radiation-Induced Xerostomia
Keywords: Xerostomia; Radiotherapy of head and neck; BioXtra
MeSH Terms: conditions — Xerostomia | interventions — BioXtra

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bioxtra spray and mouth rinse (Other): Drug: BioXtra spray or mouth rinse Patients had been xerostomia due to radiation of head and neck were selected for the study. Gender, age, medical history, VAS, dichotomous questionnaire of xerostomia , and other treatment used for this disease were recorded. Local ethical committee approval was obtained before the trial started and all patients gave written informed consent. Patients were randomly divided into two groups .First group received BioXtra spray and second group used BioXtra mouth rinse for 2 weeks and then 1 weeks wash -out period and for other 2 weeks drugs is switched . Each patients was examined at the beginning of the therapy ,and then 2 weeks after therapy and 35 days after first visit.
  Interventions: Drug: bioxtra

INTERVENTIONS:
Drug: bioxtra — spray /mouth rinse
  Other Names: saliva subsitute

SUMMARY:
The present study compared the efficacy of BioXtra spray and mouth rinse in the relief of radiotherapy-induced xerostomia in patients referred to Cancer Institute, Tehran Imam Khomeini Hospital.

DETAILED DESCRIPTION:
Xerostomia or dry mouth is an important complication of radiotherapy for head and neck regions producing serious discomfort for patients with a significant reduction in their quality of life. Symptomatic treatments for the disease include maintain oral hygiene and use of artificial saliva substitutes.

Due to limited studies on efficacy compounds BioXtra, present study compared the effects of spray and mouth rinse BioXtra in symptoms of xerostomia in patients under head and neck cancer radiotherapy .

ELIGIBILITY:
Inclusion Criteria:

* complaint of xerostomia after head and neck radiotherapy
* patient must have given written informed consent

Exclusion Criteria:

* age under 18 years
* history of any treatment for cancer in the last 3 months
* recurrence of cancer and end stage of it
* diabetes mellitus
* sjogren syndrome or other medical causes of xerostomia
* drug therapy which might induce xerostomia
* refusal of cooperation or consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
improvement of xerostomia | 2 weeks
  change of symptoms of xerostomia is measured by Visual Analogue Scale and Dichotomos questionnaire[ Time Frame: baseline compared with measures on day 14

SECONDARY OUTCOMES:
comparative analysis of improvement xerostomia between 2 drugs | 5 weeks
  change of symptoms of xerostomia is measured by Visual Analogue Scale and Dichotomos questionnaire[ Time Frame: baseline compared with measures on day 35 and comparative analysis between BioXtra spray and mouth rinse

CONTACTS AND LOCATIONS:
Overall Officials: Mahin Bakhshi, DDS/MS, Study Chair — Qazvin University Of Medical Sciences; Touba Karagah, DDS, Principal Investigator — QUMS; Soheila Manifar, DDS/MS, Study Director — Imam Khomeini Hospital; Navid Mohamadi, PHD, Study Director — QUMS; Abbas Hosseinmardi, DDS, Principal Investigator — QUMS
Locations (1):
- Qazvin University of Medical Sciences, Qazvin, Qazvin Province, Iran